CLINICAL TRIAL: NCT05830084
Title: Phase Ib Study of the Combination of Regorafenib With Conventional Chemotherapy for the Treatment of Newly Diagnosed Patients With Multimetastatic Ewing Sarcoma
Brief Title: Phase Ib / Regorafenib With Conventional Chemotherapy/Newly Diagnosed Patients/ Multimetastatic Ewing Sarcoma
Acronym: REGO-INTER-EWI
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-002874-10; 2023-503322-39-00 (EU CTIS Number); 2022/3545 (Other: CSET number)
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — regorafenib

STUDY DESIGN:
Intervention Model Description: Patient with Ewing Sarcoma male or female age ≥2 years and <50 years (from second birthday to 49 years 364 days) who are assessed as medically fit to receive the Ewing sarcoma standard multimodal treatment and regorafenib. Patients will benefit from the social security coverage in force in their country and will have received free and informed information allowing the collection of their consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction chemotherapy (VDC/IE) and local treatment /consolidation chemotherapy (Experimental): Standard ES treatment consists of: induction chemotherapy (VDC/IE) and local treatment (surgery/radiotherapy), followed by consolidation chemotherapy (VC/IE)/ Bu-Mel (according to physician and patient choice).
  Regorafenib will be administered during induction chemotherapy (VDC/IE) and during consolidation chemotherapy with conventional chemotherapy (VC/IE) but not Bu-Mel therapy Conventional chemotherapy will be administered at the recommended dose (100%) and only regorafenib will be escalated/de-escalated.
  Regorafenib will only be given concomitant to radiotherapy in case the primary tumor is located in the extremities. In case of primary tumors located in the pelvis, abdomen, thorax, spine, brain, head or neck, regorafenib will be stopped at least 1 week before start of radiotherapy.
  Interventions: Drug: regorafenib tablet

INTERVENTIONS:
Drug: regorafenib tablet — Regorafenib will be escalated/de-escalated, starting at DL0:
  * DL1: 82 mg/m^2 once daily for 21 days/28 days (max 160mg) (100% of the RP2D)
  * DL0 (starting dose): 66 mg/m^2 once daily for 21 days/28 days (max 120mg) (80% of the RP2D)
  * DL-1: 50 mg/m^2 once daily for 21 days/28 days (max 80mg) (60% of the RP2D)

SUMMARY:
New drug efficacy in ES has been disappointing in the last decades and no new drugs have been successfully introduced up to now in front line treatment. Among the tested drugs, early clinical data suggest that strategies using multi-targeted tyrosine kinase inhibitors (TKI) with anti-angiogenic activities are among the most efficient and may be beneficial in the treatment of patients with ES.

Several TKI have been and are currently being tested as single-agent in patients with relapsed/refractory ES with encouraging results in phase II trials. Regorafenib has shown promising activity in Ewing sarcoma relapse setting, Nevertheless, regorafenib has never been combined with the intensive chemotherapy VDC/IE schedule and therefore this combination needs to be evaluated in order to avoid dose reduction of the current standard treatment and hence its efficacy.

The current clinical trial has been therefore designed to test the feasibility of regorafenib with ES conventional chemotherapy. It consists of a phase Ib that will only recruit patients with multi-metastatic (other than lungs/pleura only) ES, that present the highest unmet medical need (2 year EFS: 33%, similar to patients with relapse/refractory ES).

DETAILED DESCRIPTION:
All included patients will receive standard Ewing sarcoma (ES) treatment concomitant with regorafenib.

Standard ES treatment consists of: induction chemotherapy (VDC/IE) and local treatment (surgery/radiotherapy), followed by consolidation chemotherapy (VC/IE)/ Bu-Mel (according to physician and patient choice).

Regorafenib will be administered during induction chemotherapy (VDC/IE) and during consolidation chemotherapy with conventional chemotherapy (VC/IE) but not Bu-Mel therapy

Conventional chemotherapy will be administered at the recommended dose (100%) and only regorafenib will be escalated/de-escalated, starting at DL0:

* DL1: 82 mg/m^2 once daily for 21 days/28 days (max 160mg) (100% of the RP2D)
* DL0 (starting dose): 66 mg/m^2 once daily for 21 days/28 days (max 120mg) (80% of the RP2D)
* DL-1: 50 mg/m^2 once daily for 21 days/28 days (max 80mg) (60% of the RP2D) Regorafenib will be stopped 2 weeks before planned surgery of the primary tumor and reintroduced when adequate wound healing is obtained, concomitant with consolidation VC/IE chemotherapy.

Regorafenib will only be given concomitant to radiotherapy in case the primary tumor is located in the extremities. In case of primary tumors located in the pelvis, abdomen, thorax, spine, brain, head or neck, regorafenib will be stopped at least 1 week before start of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Any histologically and genetically confirmed Ewing sarcoma of bone or soft tissue, or round cell sarcomas which are 'Ewing's-like' but negative for EWSR1 gene rearrangement
2. Metastatic disease
3. Age ≥2 years and <50 years (from second birthday to 49 years 364 days)
4. Patient assessed as medically fit to receive the Ewing sarcoma standard multimodal treatment and regorafenib, including:

   * Absolute Neutrophil Count (ANC) ≥ 0.75x10^9/L, platelets ≥ 75x10^9/L.
   * Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 5×ULN
   * Bilirubin ≤ 2×ULN
   * Creatinine < 2x ULN or creatinine clearance >60 ml/min/1.73 m^2
   * International normalized ratio (INR)/ Partial thromboplastin time (PTT). INR and PTT ≤ 1.5 x ULN. INR & PTT ≤ 1.5xULN
5. Adequate cardiac function as evidenced by left ventricular ejection fraction (LVEF) ≥50%) at baseline, as determined by echocardiography
6. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as: a BP <95th percentile for sex, age, and height at screening (as per National Heart Lung and Blood Institute [NHLBI] guidelines) and no change in antihypertensive medications within 1 week prior to Cycle 1 Day 1. Patients >18 years old should have BP ≤ 150/90 mmHg.
7. No prior treatment for Ewing sarcoma other than surgery
8. Negative pregnancy test for female patients of childbearing potential within 7 days prior to study registration.
9. Patient agrees to use highly effective contraception during therapy and for 12 months after last trial treatment (females) or 6 months after last trial treatment (males), where applicable
10. Subject must be able to swallow and retain oral medication.
11. Written informed consent from the patient and/or the parent/legal guardian, according to local, regional or national regulation prior to any study specific procedures.
12. Patients must be affiliated to a social security system or beneficiary of the same, as per local regulatory requirements (France only)

Exclusion Criteria:

1. Localized tumor or metastatic disease to lung/pleura only.
2. Contra-indication to the Ewing sarcoma standard multimodal treatment
3. Pregnant or breastfeeding women or intending to become pregnant during the study.
4. Follow-up not possible due to social, geographic or psychological reasons
5. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter absorption of oral drugs
6. A clinically significant ECG abnormality, including a marked prolonged QTcF interval (eg, a repeated demonstration of a QTcF interval >480 msec) Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality, unstable angina, active coronary artery disease and myocardial infarction within 6 months before randomization.) Uncontrolled hypertension (systolic pressure >150 mmHg or diastolic pressure > 90 mmHg on repeated measurement) despite optimal medical management
7. Previous arterial or venous thromboembolisms Grade ≥ 3 per CTCAE v5.0
8. Hypersensitivity to any active substance or to any excipients
9. Radiographic evidence of encasement or invasion of a major blood vessel or of intratumoral cavitation
10. Major surgical procedure or significant traumatic injury within 28 days before starting study treatment
11. Non-healing wound, ulcer or bone fracture.
12. Uncontrolled systemic or local infection requiring systemic treatment
13. Any anticoagulant therapy (risk of hemorrhage with Regorafenib)
14. Interstitial lung disease with ongoing signs and symptoms.
15. Known prior history of HBV, HCV, HIV
16. Any other medical or other condition that, in the opinion of the investigator(s), would preclude the subject's participation in this clinical study

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose-Limiting Toxicities (DLT) | 28 days after the start of treatment
  The dose-finding escalation will be driven by the occurrence of Dose-Limiting Toxicities (DLT), assessed over the first 28-day cycle (cycle 1), and defined as any of the following haematological and non-haematological events that occur during the DLT period (4 weeks after the start of treatment = cycle 1) and are at least possibly related (possibly, probably, or definitely) attributable to VDC/IE + regorafenib:
  * Any cardiac toxicity grade ≥ 3
  * Any grade 3 or 4 (hematological or non-hematological) toxicity leading to delay of start of next course by > 7 days (i.e: starting > day 21).
  * Any dose interruption or reduction due to toxicity which results in administration of less than 80% of the planned dosage of regorafenib or 75% of the planned dosage of chemotherapy.
  * Any grade 3 or 4 toxicity resulting in discontinuation of the new combination
  * Any grade 5 toxicity related to study treatment (death)

SECONDARY OUTCOMES:
Overall Survival (OS) | Until 18 months after inclusion of the last patient
  Defined as the time from start of anti-cancer treatment to death, irrespective of the cause. Surviving patients will be censored at their last follow-up date
Progression-Free Survival (PFS) | Until 18 months after inclusion of the last patient
  Defined as the time from start of anti-cancer treatment to first event, where an event is progression without complete remission, recurrence following complete remission or death.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Berlanga, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (13):
- Australia (4):
  - Queensland Children's Hospital, Brisbane
  - Monash Children's Hospital, Clayton
  - Royal Children's Hospital, Parkville
  - Perth Children's Hospital, Perth
- Rigshospitalet, Copenhagen, Denmark
- France (5):
  - CHU Bordeaux, Bordeaux
  - Centre Oscar Lambret, Lille
  - centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Gustave Roussy, Villejuif, Île-de-France Region
- Istituto Nazionale dei Tumori, Milan, Italy
- Princess Máxima Center, Utrecht, Netherlands
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No